CLINICAL TRIAL: NCT03419936
Title: Distribution of Helicobacter Pylori in Remnant Stomach After Subtotal Gastrectomy
Brief Title: Distribution of Helicobacter Pylori After Gastrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Yong Ahn, Associate professor, Asan Medical Center
Other Study IDs: 2015-0823
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Helicobacter Pylori Infections
Keywords: Stomach Neoplasms; Helicobacter pylori; Subtotal gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Endoscopic biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Helicobacter pylori(HP) positive: Participants who are diagnosed with gastric cancer and Helicobacter Pylori infection will be treated with subtotal gastrectomy.
  Interventions: Diagnostic Test: Endoscopic biopsy

INTERVENTIONS:
Diagnostic Test: Endoscopic biopsy — 1. Pre-operation (initial diagnosis) Assessment atrophy and metaplasia in stomach, Check Helicobacter pylori
  2. Post-subtotal gastrectomy (After 6 months) Assess the distribution of helicobacter pylori after subtotal gastrectomy.
  3. Post-subtotal gastrectomy (After 12 months) Assess the distribution of helicobacter pylori after subtotal gastrectomy.
  4. Post-subtotal gastrectomy (After 24 months) Assess the distribution of helicobacter pylori after subtotal gastrectomy.

SUMMARY:
The purpose of this study is to know the distribution of Helicobacter pylori in stomach before subtotal gastrectomy and after subtotal gastrectomy.

DETAILED DESCRIPTION:
Endoscopy and biopsy will be performed to investigate the distribution of Helicobacter pylori before and after subtotal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are indicated to subtotal gastrectomy due to gastric neoplasm
2. Aged between 19 to 75 years
3. Informed consent

Exclusion Criteria:

1. Previous history of Helicobacter pylori eradication
2. Previous history of proton pump inhibitor use within 6 months

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size will be determined based on the analysis the distribution rate of Helicobacter pylori at first 60 patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-03-21 (Actual); Primary Completion 2020-03-21 (Estimated); Study Completion 2020-03-21 (Estimated)

PRIMARY OUTCOMES:
Distribution of Helicobacter Pylori After Gastrectomy | Change in the distribution of Helicobacter Pylori at 2 years
  Analysis the change of Helicobacter pylori according to the subtotal gastrectomy

SECONDARY OUTCOMES:
Change of atrophy after gastrectomy | Change in the atrophic status at 2 years
  Analysis the change of atrophic status according to the subtotal gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ji Yong Ahn, Professor, Principal Investigator — Study Principal Investigator Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No